CLINICAL TRIAL: NCT02584608
Title: Phase 2a Study of Interferon Gamma-1b for the Treatment of Autosomal Dominant Type 2 Osteopetrosis
Brief Title: Use of ACTIMMUNE in Patients With ADO2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Horizon Pharma Ireland, Ltd., Dublin Ireland (Industry)
Responsible Party: Principal Investigator, Michael Econs, MD, Professor of Endocrinlogy and Metabolism, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1510340687
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Autosomal Dominant Osteopetrosis Type 2
MeSH Terms: conditions — Osteopetrosis | interventions — interferon gamma-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): ACTIMMUNE 50 µg/m2 subcutaneously three times per week (TIW) for 8 weeks
  Interventions: Drug: ACTIMMUNE

INTERVENTIONS:
Drug: ACTIMMUNE

SUMMARY:
This study is an open label use of ACTIMMUNE for patients with Autosomal Dominant Osteopetrosis Type 2(ADO2). Effects of treatment will be evaluated after 14 weeks on ACTIMMUNE by bone resorption markers. This study will treat 12 patients with ADO2 recruited from Indiana University and Riley Hospital for Children at Indiana University Health.

DETAILED DESCRIPTION:
This is a single center, open-label, dose-escalation study evaluating the efficacy, as defined by biochemical endpoints, and safety profiles of ACTIMMUNE in ADO2 subject.

The investigators will treat 12 ADO2 subjects (children or adults age 3-65) with Actimmune® via a dose escalation protocol to a dose of 50 µg/m2 subcutaneously three times per week (TIW) for 8 weeks. If serum CTX does not increase by more than 25% by week 8, the dose will be increased to 100 µg/m2 subcutaneously TIW.

Individual subjects in whom ACTIMMUNE administration increases bone resorption markers during the 14 weeks of this trial will be eligible for a 1 year extension trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is diagnosed with clinically significant ADO2 as determined by the investigator.

   Individuals will be screened who have either been diagnosed with osteopetrosis and have a clinical phenotype and/or family history that is consistent with ADO2, have been told that they have an abnormally high bone density (>3SD above mean for age and sex), or a clinical presentation consistent with ADO2. Initial contact will be with members of ADO2 kindreds who have known disease.
2. Provide written informed consent for competent adults and for minors provide written assent (if appropriate) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures
3. Ages 3 to 65 years inclusive.
4. Willing to use reliable method of contraception [i.e. oral or patch hormonal contraceptives, intrauterine device, physical barrier methods, tubal ligation or hysterectomy, vasectomy (partner) or abstinence] throughout the study and for 30 days after the last dose of study drug.

Exclusion Criteria:

1. Any unstable illness that in the investigator's opinion precludes participation in the study.
2. Serum calcium >10.6 mg/dl at screening.
3. eGFR using the MDRD equation in adults (or the modified Schwartz equation for children) of < 35 ml/min/1.73m2.
4. Nephrocalcinosis on screening ultrasound Grade 3 or higher [18]. Subjects with grade 3 or higher nephrocalcinosis will be excluded because we anticipate that use of study drug will increase bone resorption, resulting in increased urinary calcium excretion, which could, potentially, lead to worsening nephrocalcinosis. The grading scale is listed below:

0 = Normal

1. = Faint hyperechogenic rim around the sides and tip of the medullary pyramids
2. = More intense echogenic rim with echoes faintly filling the entire medullary pyramid
3. = Intense echoes throughout the medullary pyramid
4. = Solitary focus of echoes at the tip of the medullary pyramid/nephrolithiasis

5. Use of any investigational product (drug or device) within 30 days prior to randomization.

6. Subject reported history of hepatitis C.

7. A recent (past 5 years) history of alcoholism or intravenous drug abuse.

8. History of hypersensitivity to IFN-ɣ or E. coli-derived products.

9. History of liver disease as evidenced by laboratory results at Screening (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] >2x the upper limit of normal), except when in the opinion of the investigator the liver disease is caused by extra medullary hematopoiesis.

10. Pregnant or nursing women or those who plan on becoming pregnant during the study.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Econs, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Imel EA, Liu Z, Acton D, Coffman M, Gebregziabher N, Tong Y, Econs MJ. Interferon Gamma-1b Does Not Increase Markers of Bone Resorption in Autosomal Dominant Osteopetrosis. J Bone Miner Res. 2019 Aug;34(8):1436-1445. doi: 10.1002/jbmr.3715. Epub 2019 May 13. PMID 30889272

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: ACTIMMUNE 50 µg/m2 subcutaneously three times per week (TIW) for 8 weeks
  ACTIMMUNE
Period: Overall Study
Arm/Group | Treatment
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: Total matches.
  years
    Total | 30.48 [8.1 to 50.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Changes in Bone Resorption Markers From Baseline to 14 Weeks.
Description: Evaluate for changes in bone resorption markers including CTX, NTX/creatinine ratio between baseline and 14 weeks
Time Frame: baseline, 14 weeks
Population: All subjects
Measure: Mean (Full Range); unit: percentage of change
Arm/Group | Treatment
Number analyzed (Participants) | 12
percentage of change
  Percent change of CTX | 2.2 [-35.7 to 90.5]
  Percent change of NTX/creatinine ratio | -2.1 [-50.5 to 55.5]

2. Secondary Outcome: Change in Bone Turnover Markers Between After Completion of 6-12 Weeks of Treatment
Description: Evaluate for changes in bone turnover markers including TRAP5b, NTX, CTX/TRAP5b ratio after 6-12 weeks of treatment.
Time Frame: 6-12 weeks
Population: all subjects
Measure: Mean (Full Range); unit: percentage of change
Arm/Group | Treatment
Number analyzed (Participants) | 12
percentage of change
  TRAP5B | -15.34 [-57.07 to 13.1]
  NTX | -2.09 [-50.51 to 55.54]
  CTX/TRAP5b ratio | 26.31 [-35.91 to 144.57]

ADVERSE EVENTS:
Time Frame: From signing consent till final followup at 18 weeks (4 weeks after stopping study drug)
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 10/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=12)
Headache (Nervous system disorders) | 10
Fatigue (Nervous system disorders) | 9
nausea (Gastrointestinal disorders) | 9
flu like symptoms (Product Issues) | 8
myalgia (Musculoskeletal and connective tissue disorders) | 7
white blood cell decreased (Blood and lymphatic system disorders) | 6
arthralgia (Musculoskeletal and connective tissue disorders) | 5
diarrhea (Gastrointestinal disorders) | 5
neutrophil count decreased (Blood and lymphatic system disorders) | 5
vomiting (Gastrointestinal disorders) | 5
back pain (Musculoskeletal and connective tissue disorders) | 4
injection site reaction (Skin and subcutaneous tissue disorders) | 4
pain in extremity (Musculoskeletal and connective tissue disorders) | 4
bone pain (Musculoskeletal and connective tissue disorders) | 4
chills (Immune system disorders) | 3
CPK increased (Investigations) | 3
hypertriglycerides (Endocrine disorders) | 3
platelet count decrease (Blood and lymphatic system disorders) | 3
anemia (Blood and lymphatic system disorders) | 2
constipation (Gastrointestinal disorders) | 2
dizziness (Nervous system disorders) | 2
agitation (Psychiatric disorders) | 1
aspartate Aminotransferase increased (Blood and lymphatic system disorders) | 1
chest wall pain (Musculoskeletal and connective tissue disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT02584608/Prot_SAP_000.pdf